CLINICAL TRIAL: NCT06251895
Title: Association of the Systemic Immune-inflammation Index (SII) and Severity of Diabetic Ketoacidosis in Patients With Type 1 Diabetes Mellitus: A Retrospective Cohort Study
Brief Title: Association of Systemic Immune-inflammation Index and Severity of Diabetic Ketoacidosis in Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Jahra Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Aon, Principal Investigator, Jahra Hospital
Other Study IDs: J1 - 18072023
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Ketoacidosis
Keywords: Complete blood count; diabetes mellitus; diabetic ketoacidosis; systemic immune inflammation index.
MeSH Terms: conditions — Diabetic Ketoacidosis; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild DKA: pH < 7.3 or serum bicarbonate <18 mmol/L
  Interventions: Other: DKA protocol
- moderate DKA: pH < 7.2 or serum bicarbonate <10 mmol/L
  Interventions: Other: DKA protocol
- severe DKA: pH < 7.1 or serum bicarbonate <5 mmol/L
  Interventions: Other: DKA protocol

INTERVENTIONS:
Other: DKA protocol — IV fluids and IV insulin as per guidelines. reference 1-2

SUMMARY:
Diabetic ketoacidosis (DKA) is the most serious metabolic complication of type 1 diabetes mellitus (T1DM). Insulin deficiency and inflammation play a role in the pathogenesis of DKA. The investigators aim to assess the systemic immune-inflammation index (SII) as a marker of severity among T1DM patients with DKA and without infection.

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is one of the most severe acute metabolic complications of diabetes mellitus (DM). Therefore, DKA patients require prompt treatment and any delay in identifying severe DKA cases can lead to worse outcomes. DKA provokes a systemic inflammatory response through increased levels of various cytokines such as interleukin (IL)-8, IL-6, IL-10, tumor necrosis factor-alpha (TNF-α), and IL-1B. This will lead to cellular activation, cellular adhesion, increased oxidative stress, and endothelial damage, possibly contributing to complications. Consequently, surrogate markers of inflammation and immune status may help in the early identification of patients with severe DKA.

The systemic immune-inflammation index (SII) had a better prognostic value compared to NLR and PLR among cancer patients. Recently, studies have suggested a link between SII and increased risk of atherosclerotic cardiovascular disease (ASCVD), hepatic steatosis, and worse outcomes among hypertensive patients and patients with stroke.

Therefore, the investigators aim to examine SII as a marker of severity in T1DM patients with DKA in an uninfected state.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T1DM
* Hospitalization because of DKA
* Age ≥ 12 years.

Exclusion Criteria:

* Diagnosis of T2DM
* Diagnosis of Infection
* Renal impairment
* Malignancy
* ASCVD (atherosclerotic cardiovascular disease)
* History of any medical condition or medications that can change CBC parameters or cause metabolic acidosis
* Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 DM hospitalized because of DKA.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
SII | Day 1 (baseline)
  SII = (neutrophil × platelet) / lymphocyte.

SECONDARY OUTCOMES:
ICU admission | Hospital stay up to one week
  need for ICU admission
readmission | within 90 days
  readmission because of DKA

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED AON, PHD, Principal Investigator — Cairo University
Locations (1):
- Jahra Hospital, Kuwait, Al Jahra Governorate, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided
Datasets analyzed during the current study will be available upon reasonable request from the corresponding author and after IRB approval.

REFERENCES:
- [Background] Dhatariya KK; Joint British Diabetes Societies for Inpatient Care. The management of diabetic ketoacidosis in adults-An updated guideline from the Joint British Diabetes Society for Inpatient Care. Diabet Med. 2022 Jun;39(6):e14788. doi: 10.1111/dme.14788. Epub 2022 Feb 27. PMID 35224769
- [Background] Glaser N, Fritsch M, Priyambada L, Rewers A, Cherubini V, Estrada S, Wolfsdorf JI, Codner E. ISPAD clinical practice consensus guidelines 2022: Diabetic ketoacidosis and hyperglycemic hyperosmolar state. Pediatr Diabetes. 2022 Nov;23(7):835-856. doi: 10.1111/pedi.13406. No abstract available. PMID 36250645